CLINICAL TRIAL: NCT00873392
Title: Efficacy of Transdermal Nicotine, on Motor Symptoms in Advanced Parkinson's Disease(One Daily Administration).A Controlled Randomised Study, in Two Parallel Groups and Single Blind in 40 Patients.
Brief Title: Efficacy of Transdermal Nicotine, on Motor Symptoms in Advanced Parkinson's Disease
Acronym: NICOPARK2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P 051031
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Parkinson's disease; Motor fluctuation; Nicotine; Drug treatment; neuroprotection
MeSH Terms: conditions — Parkinson Disease | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Experimental drug
  Interventions: Drug: Transdermal nicotine
- 2 (Active Comparator): Usual treatment
  Interventions: Other: Usual drug treatment of Parkinson's disease

INTERVENTIONS:
Drug: Transdermal nicotine — Steps of 5 mg until 20 mg Then steps of 10 mg until the dose of 90mg or the maximal tolerated dose One stable dose phase, (90 mg or maximal tolerated dose) during 28 weeks
  Arms: 1
Other: Usual drug treatment of Parkinson's disease — Usual drug treatment of Parkinson's disease
  Arms: 2

SUMMARY:
Medical treatment of idiopathic Parkinson disease motor symptoms requires dopaminergic drugs, with long term disabling side effects. (fluctuations, dyskinesia, ON/OFF phenomena). Use of nicotine in Parkinson's disease has been suggested by the lowest prevalence of smokers among Parkinsonian patients. However, controlled studies provided conflicting results. One of our patients showed a substantial decrease of his parkinsonian symptoms under transdermal nicotine-therapy. Currently, this patient has been treated since 8 years with an excellent safety, especially on cardiovascular level. Otherwise, the investigators performed an open pilot safety and feasibility study in 6 patients, which demonstrated the possibility of a controlled study. In this study, all patients received daily doses during several months until 105 mg/day and could, in parallel, decrease their L-Dopa and agonists doses, improving their motor scores.

The investigators now propose a phase II, controlled, single blind and randomised efficacy study (n=40) in 2 parallel groups. (1 group transdermal nicotine-therapy / 1 control group without additional therapy) The main objective is to verify the correlation between UPDRS (score III) motor score and the administrated nicotine dose. This study will also allow the evaluation of nicotine neuroprotective effect. The incrementation phase by weekly steps of 5 mg until 20 mg, then 10 mg to reach 90 mg/j or the maximal tolerated dose, will last on 11 weeks and will be followed by a 28 weeks phase at this stable dose. After this maximal dose "plateau phase", treatment will be progressively decreased by 15 mg weekly steps, over a de 6-week period followed by a five-week wash out phase.

Taking into account results from the pilot study, a long-term high doses treatment, seems to be liable to improve patients who deeply suffer from their disease. This is why the investigators now propose this monocentric institutional project.

DETAILED DESCRIPTION:
Experimental plan

Phase II controled study, in 40 patients, randomised in single blind, and in 2 groups:

* One group treated by transdermal nicotine-therapy (N= 20),
* One group without additional therapy (N= 20).

This study will consist in :

* One phase of weekly incrementations of dose during 11 weeks,

  * Steps of 5 mg until 20 mg
  * Then steps of 10 mg until the dose of 90mg or the maximal tolerated dose
* One stable dose phase, (90 mg or maximal tolerated dose) during 28 weeks,
* One phase of decrementing: treatment will be progressively decreased in a 6 weeks period,

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic Parkinson's disease according to the United Kingdom Parkinson's Disease Society Brain Bank (UKPDSBB), since at least three years,or treated by L-dopa for 2 years minimum with motor fluctuations (amendment 12/10/2010)
* Patients aged between 35 and 70 years inclusive,
* L-Dopa responders: L-Dopa test with an improvement of over 30 % of UPDRS-III motor score,
* L-Dopa treatment since at least three years,
* Patients with Parkinson's disease stage maximum IV ("OFF" state) according to the modified Hoehn and Yahr classification (without treatment since at least 12 hours), and III maximum in "ON" state,
* Non smoker,
* Signed Informed Consent

Exclusion Criteria:

* Previous neurosurgery for Parkinson's disease,
* Weight < 45 kg or > 100 kg,
* Previous Parkinson's disease treatment by transdermal nicotine-therapy discontinued less than 6 months before inclusion,
* History of allergy to Nicotine,
* History of allergy to transdermal device,
* Cutaneous disorders wich could disturb use of transdermal device,
* Cognitive disorders, (Mattis score < 125)
* History or detection at inclusion of cardiac arrhythmia,
* History of coronary failure,
* History of cardiac failure, (NYHA from II to IV & ejection fraction (EF) < 40%)
* Severe arterial hypertension (diastolic > 100 mmHg) or uncontrolled,
* Symptomatic orthostatic hypotension, (2 points of differential in standing position and systolic <100mm Hg or clinical evidence)
* History of stroke or occlusive peripheral vascular disease,
* History of hyperthyroid,
* History or detection at inclusion of type I or II diabetes, (HbA1c < 11%)
* History of pulmonary disease: asthma, chronic obstructive pulmonary disease (COPD),
* History of auto-immune disease,
* Progressive depression, suicide attack, acute psychosis, invasive hallucinations, psychiatrist opinion harmful for a correct compliance to experimentation,
* History or recent gastroduodenal ulcer, (< 3 months)
* History or detection at inclusion of hepatobiliary or renal failure, (clearance< 60 mL/min)
* Pregnancy, breast-feeding,
* Absence of effective contraception in women in childbearing potential,
* Treatment by nifedipine, beta-blockers, diuretics, insulin and H2 antihistaminics for potential side effects in combination with nicotine,
* Patients unlikely to be compliant or to fully cooperate during the study.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-02; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Comparison of motor scores in defined off condition : UPDRS III motor score assessed in "defined OFF" condition in comparison with control group. | after 20/39 weeks of treatment at maximal administered dose of nicotine

SECONDARY OUTCOMES:
Evaluation of UPDRS III motor score assessed in "defined OFF" condition | after 20 weeks of treatment in comparison with control group
Improvement of UPDRS III motor score assessed in "defined ON" condition | after a 12 hours discontinuation of antiparkinsonian treatments after 11, 20 and 39 weeks of treatment
Evaluation of motor benefit (UPDRS "OFF" and "ON") | after a 28 weeks treatment period at stable dose of 90 mg
Evaluation of neuroprotection, (SPECT DaTSCAN and UPDRS "OFF") | after 5 weeks of study treatment discontinuation
Persistence of motor benefit (UPDRS "OFF" and "ON") | after 5 weeks of study treatment discontinuation
Decrease of total daily L-Dopa dose (or calculated equivalent in case of polytherapy) | after 20 and 39 weeks of treatment
Improvement of quality of life (ADL and PDQ 39 scales) | after 20 and 39 weeks of treatment
Decrease of daily percentage of "OFF" phase | after 20 and 39 weeks of treatment
Improvement of dyskinesia score, (UPDRS IV) | during the study
Relation dose / effect of nicotine | end of the study
Estimation of the most effective and tolerated dose of nicotine per kg | end of the study
Improvement of cognitive functions assessed by Mattis scale | after 39 weeks of treatment
Comparison of all parameters between the 2 groups of patients | after study treatment discontinuation, (Week 50)
Compliance to nicotine treatment | during treatment
Tolerance of transdermal nicotine | during the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pierre CESARO, PUPH, Principal Investigator — Groupe Hospitalier Albert Chenevier Henri Mondor
Locations (1):
- Groupe Hospitalier Albert Chenevier Henri Mondor, Créteil, France

REFERENCES:
- [Result] Villafane G, Cesaro P, Rialland A, Baloul S, Azimi S, Bourdet C, Le Houezec J, Macquin-Mavier I, Maison P. Chronic high dose transdermal nicotine in Parkinson's disease: an open trial. Eur J Neurol. 2007 Dec;14(12):1313-6. doi: 10.1111/j.1468-1331.2007.01949.x. Epub 2007 Oct 17. PMID 17941858